CLINICAL TRIAL: NCT04719767
Title: Application of Visual Laryngeal Mask Airway Combined With Endotracheal Intubation in Non-head and Neck Surgery Under General Anesthesia
Brief Title: Application of Visual Laryngeal Mask Airway Combined With Endotracheal Intubation in General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Xia Ruan, Attending doctor of the Department of Anesthesiology, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PUMCH-rx
Record Dates: First submitted 2021-01-06; First posted 2021-01-22 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: General Anesthesia; Laryngeal Mask; Endotracheal Intubation; Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patients, surgeons and the ones who collect data will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- visual (Experimental): In the visual group, a visual laryngeal mask was placed and endotracheal intubation was guided under visual conditions. The endotracheal tube was removed 10 minutes before the end of the operation, and the laryngeal mask was retained.
  Interventions: Device: visual laryngeal mask
- Non-visual (No Intervention): In the non-visual group, laryngeal mask airway was inserted. After clinical judgment of good counterpoint, endotracheal intubation was inserted blindly through LMA. Endotracheal intubation was removed 10 minutes before the end of the operation, and the laryngeal mask airway was retained.

INTERVENTIONS:
Device: visual laryngeal mask — After anesthesia induction, visual laryngeal mask airway was placed in the visual group and tracheal intubation was guided under visual conditions. In the non-visual group, laryngeal mask airway was inserted, after clinical judgment of good counterpoint of the laryngeal mask, endotracheal intubation was inserted blindly through LMA. Selection of laryngeal mask airway (LMA) model: the ideal body weight of the patient was calculated.
  Arms: visual

SUMMARY:
To study the advantages of visual laryngeal mask combined with endotracheal intubation in general anesthesia surgery, we compared intubation time, intubation times and intubation success rate of endotracheal intubation through laryngeal mask airway under visual and non-visual conditions, at the same time, the laryngeal mask displacement rate, volume of secretion in airway, the incidence of laryngeal spasm, the incidence and severity of postoperative oropharyngeal pain were also compared between two groups.

DETAILED DESCRIPTION:
After entering the operating room, the patient received routine general anaesthesia monitoring, and anesthesia induction was conducted after three-party verification. Propofol (plasma target-controlled concentration: 3.5ug/ mL), midazolam (0.05mg/kg), fentanyl (2ug/kg) and rocuronium (0.6mg/kg) were used to induce the drugs.

After anesthesia induction, visual laryngeal mask airway was placed in the visual group and endotracheal intubation was guided under visual conditions. In the non-visual group, after judging the position of laryngeal mask by clinical experience, endotracheal intubation was inserted blindly. Selection of laryngeal mask airway (LMA) model based on: the ideal body weight of the patient, 3 was selected for the body weight of 30-50kg, 4 for the body weight of 50-70kg and 5 for the body weight > 70kg. The endotracheal tube intubation time, intubation times and intubation success rate of the two groups were recorded.

During the operation, propofol and fentanyl are used for anesthesia maintenance, and the anesthesiologist adjusts the anesthesia depth according to his/her own experience. Ten minutes before the end of the operation, endotracheal intubation was removed and the laryngeal mask airway was retained. The displacement rate of the laryngeal mask airway, the volume of secretion in airway and the incidence of laryngeal spasm were compared between the two groups.

After the surgery, the residual muscle relaxation was antagonized, and the laryngeal mask was removed after the patient regained consciousness and reached the extubation criteria. The hemodynamic parameters and the severity of cough during laryngeal mask airway removal were recorded. The incidence and severity of oropharyngeal pain, oropharyngeal numbness, hoarseness, nausea, and vomiting were assessed immediately after the patient woke up and was followed up before leaving the recovery room and on the first day after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70
* American Society of Anesthesiologist physical status (ASA) Ⅰ-II
* Undergoing non-head and neck surgery under general anesthesia with endotracheal intubation
* Sign the informed consent voluntarily;

Exclusion Criteria:

* Not willing to participate in the study or not able to sign the informed consent
* American Society of Anesthesiologist physical status (ASA) Ⅲ-Ⅳ
* Weight <30kg or BMI>40 kg/m2
* High risk of reflux aspiration
* Combined with severe respiratory disease
* Combined oropharyngeal lesions affect the laryngeal mask insertion
* Oropharyngeal pain in the last two weeks.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Intubation time (second) | intraoperative
  Compare the time of endotracheal intubation through laryngeal mask airway under visual and non-visual conditions

SECONDARY OUTCOMES:
Success rate of the endotracheal intubation (%) | intraoperative
  Compare success rate of endotracheal intubation through laryngeal mask airway under visual and non-visual conditions
Displacement rate of the laryngeal mask airway (%) | Immediately after operation
  Compare displacement rate of the laryngeal mask airway after tracheal intubation removal under visual and non-visual conditions
Incidence of oropharyngeal pain as assessed by the VAS | postoperative one day
  On the first day after operation, the patients were asked to score the oropharyngeal pain. Based on the distribution of pain VAS scores in postsurgical patients, the following cut points on the pain VAS have been recommended. No pain (0 -4 mm) Mild pain (5-44 mm) Moderate pain (45-74 mm) Severe pain (75-100 mm) The significance of the Visual Analog Scale.
Incidence and severity of hoarseness as assessed by a numerical scale | postoperative one day
  Normal = 1, weakened or hoarse = 2, unable to pronounce = 3

CONTACTS AND LOCATIONS:
Overall Officials: Yuguang Huang, M.D., Study Director — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2021-01-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT04719767/Prot_000.pdf
  • Informed Consent Form (2021-01-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT04719767/ICF_001.pdf